CLINICAL TRIAL: NCT03067805
Title: Influence of Oxytocin on Romantic Jealousy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor / Research group leader, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-12
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Sexual Infidelity; Emotional Infidelity; Jealousy
Keywords: Oxytocin effect; romantic jealousy; Arousal Rating; Jealousy Rating

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental): Oxytocin nasal spray
  Interventions: Behavioral: Sexual Infidelity Condition; Behavioral: Emotional Infidelity Condition; Behavioral: Neutral Condition; Behavioral: Player in Jealousy Condition; Behavioral: Player in Non-Jealousy Condition
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Behavioral: Sexual Infidelity Condition; Behavioral: Emotional Infidelity Condition; Behavioral: Neutral Condition; Behavioral: Player in Jealousy Condition; Behavioral: Player in Non-Jealousy Condition

INTERVENTIONS:
Behavioral: Sexual Infidelity Condition
Behavioral: Emotional Infidelity Condition
Behavioral: Neutral Condition
Behavioral: Player in Jealousy Condition
Behavioral: Player in Non-Jealousy Condition

SUMMARY:
The aim is to evoke romantic jealousy between couples and investigate whether oxytocin has effect on it.

DETAILED DESCRIPTION:
In a double-blind, between- subject placebo (PLC) controlled design,investigators plan to test the effect of intranasal oxytocin on romantic jealousy evoked by the Imaginary of Partner's Infidelity Task and Cyberball Game in romantically attached subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy couples in romantic relationship for more than 3 months and have intimate experience with each other before.

Exclusion Criteria:

* medical or psychiatric illness

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2016-02; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Arousal and jealousy ratings as assessed by Likert Scales | 145 Minutes
  Oxytocin effect on arousal and jealousy on sexual and emotional infidelity sentences

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China